CLINICAL TRIAL: NCT00840437
Title: Health Status of Patients Enrolled in the OPTions In Myocardial Ischemic Syndrome Therapy (OPTIMIST) Program
Brief Title: Quality of Life in Patients With Refractory Angina
Status: Completed | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: opt003
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Refractory Ischemia
Keywords: angina; health related quality of life
MeSH Terms: conditions — Ischemia; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The health and well being of patients with refractory angina will be assessed using validated questionnaires (SF-36 and Seattle Angina Questionnaire [SAQ]) at baseline and one year.

ELIGIBILITY:
Inclusion Criteria:

* In the OPTIMIST clinic with documented refractory angina
* Have consented to participate in the OPTIMIST Long-term Follow-up Database

Exclusion Criteria:

* Decline to participate or are unwilling to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential patients seen in the OPTions In Myocardial Ischemic Syndrome Therapy (OPTIMIST)clinic with documented refractory angina and who have consented to participate in the OPTIMIST Long-term Follow-up Database
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Health and anginal status of refractory angina patients | baseline and one year

SECONDARY OUTCOMES:
Change in Health Related Quality of Life (HRQL) | one year
Association between MACE and changes in Health Related Quality of Life (HRQL) | one year
Health Related Quality of Life (HRQL) and change in HRQL by subgroup | baseline and one year

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Henry, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- See also: Minneapolis Heart Institute Foundation — http://www.mplsheart.org/